CLINICAL TRIAL: NCT00448877
Title: Deployment of Functional Optical Brain Monitor [fNIR] in Clinical Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Jerry Levitt, MD, Drexel University College of Medicine
Organization: Drexel University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16618
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Surgical Procedures, Operative
Keywords: No specific disease is being studied, few procedures are excluded.; The focus of the study is to rule out the efficacy of the device, so the aim is to include as wide a variety of procedures as possible.

INTERVENTIONS:
Device: fNIR light emitting and sensing device

SUMMARY:
The purpose of this study is to determine whether or not a new brain function monitor can distinguish between anesthetized and awake patients. The device implemented utilizes functional near-infrared (fNIR) technology to detect anesthesia depth as well as reaction to stimuli during surgical procedure.

After obtaining consent the device is placed across the forehead of the patient. A baseline signal is obtained prior to induction. The fNIR signal is continuously recorded throughout the procedure. Key events as well as administration of drug are recorded in order to observe changes in the signal trend. Neither the device nor the light emitted is hazardous to the patient - no risks or discomforts are involved.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will have surgery
* 18-80 years old
* No restrictions on gender, race, or religion

Exclusion Criteria:

* Head and face surgery
* Induced hypotension
* Profound anemia
* Scar/tattoo on forehead
* Prior history of frontal lobe surgery
* Hemoglobinopathies
* Patients not undergoing general anesthesia
* Surgeries in the prone position
* Allergy to adhesive tape

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
This is a proof of concept study, primary outcome measure includes observation and calculation of causal relationships of oxygenated and de-oxygenated hemoglobin during administration of anesthetic.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, MD, Study Chair — Drexel University College of Medicine
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States